CLINICAL TRIAL: NCT03319069
Title: A Prospective Phase 3 Clinical Trial Of Postmastectomy Hypofractionated Radiotherapy in High Risk Breast Cancer
Brief Title: Post Mastectomy Hypofractionated Radiotherapy in High Risk Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Ahm (Other)
Responsible Party: Sponsor-Investigator, Ahmed Ahm, Dr.Hoda Hassan Mohammed Eisa, professor of clinical oncology and nuclear medicine, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17200012
Record Dates: First submitted 2017-10-02; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Intervention Model Description: Assignment Masking: open label
Masking Description: Check none
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Experimental): Hypofractionated radiotherapy women with T3-4 and /or 4 or more axillary nodes involvement post mastectomy. Hypofractionated radiotherapy 43,5 GY/15 fractions (f) /3w. to chest wall and supraclavicular nodal region.
  Interventions: Radiation: Hypofractionated radiotherapy
- group(2) (Active Comparator): Conventional fractionated radiotherapy breast cancer women with T3-4 and/ or 4 or more axillary nodes involvement post mastectomy. Conventional fractionated radiotherapy 50 Gray(GY)/25 fractions (f)/5w to chest wall and supraclavicular nodal region.
  Interventions: Radiation: Conventional fractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Hypofractionated radiotherapy 43,5 GY/15 fractions (f)/3ws. to chest wall and supraclavicular nodal region.
  .
  Arms: group (1)
Radiation: Conventional fractionated radiotherapy — 50 Gray(GY)/ 25f/5 weeks(5w) to chest wall and supraclavicular nodal region
  Arms: group(2)

SUMMARY:
The purpose of this study is to compare the efficacy and toxicities of hypofractionated radiotherapy with conventional fractionated radiotherapy in high risk breast cancer patients treated with mastectomy. It's hypothesized that the efficacy and toxicities are similar between the two groups.

DETAILED DESCRIPTION:
Eligible breast cancer patients with mastectomy and axillary dissection are divided into two groups: conventional fractionated (CF) radiotherapy of 50 Gray (GY) in 25 fractions within 5 weeks to ipsilateral chest wall and supraclavicular nodal region, and hypofractionated (HF) radiotherapy of 43.5 Gray (GY) in 15 fractions within 3 weeks to the same region. During and after radiotherapy , the patients are followed and the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Ipsilateral clinically diagnosed and histologically confirmed invasive breast cancer
* Undergone total mastectomy and axillary dissection T 3-4 and/or 4 or more positive axillary lymph nodes.
* Fit for chemotherapy ( if indicated) , endocrine therapy (if indicated), and postoperative irradiation.
* Written informed concent.
* C T3-4 , or C N2, or pathological positive axillary lymph nodes during mastectomy for patients who had received neoadjuvant chemotherapy or hormone therapy.
* No supraclavicular or internal mammary nodes metastases.
* No distant metastases .Enrollment date no more than 8 months after surgery or no more than 2 months after chemotherapy for patients who did't receive neoadjuvant therapy.
* Enrollment date no more than 2 months after surgery for patients who had received neoadjuvant systemic therapy and did't need adjuvant chemotherapy.

Exclusion Criteria:

* Patients who undergone previous irradiation to the ipsilateral chest wall and supraclavicular region
* Previous or concurrent malignant other than non melanomatous skin cancer
* Bilateral breast cancer.
* Immediate or delayed ipsilateral breast cancer reconstruction.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional control rate ipsilateral chest wall, axilla, supraclavicular and internal mammary nodal relapse. | two years
  60 female patients with high risk post mastectomy breast cancer will divided randomly into two equal groups One group will received hypofractionated (HF) regimen of postoperative radiotherapy, and group two will receive conventional fractionated (CF) regimen of postoperative local radiotherapy. in high risk breast cancer , comparison between the two treated groups.
Frequency of local recurrence. | one year
  Comparison between the treatment groups.
Toxicity outcome/ side affects that may occur with breast radiation therapy. | two years
  Comparison between the two treatment groups regarding breast irradiation toxicity outcomes and its frequency.
Histopathologic grades of the tumor. | one year
  Comparison between the two treatment groups.
Pathological tumour size (pT stage classification) | one year
  cT 3-4
Pathological node status (pN stage classification) (cN) | one year
  cN 2 (4 or more positive axillary lymph nodes.
Frequency of distant metastasis | two years
  Compare two treatment groups regarding the frequency of distant metastasis.

SECONDARY OUTCOMES:
Overall survival. | two years
  Any deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut faculty of medicine , clinical oncology and nuclear medicine department, Asyut, Egypt